CLINICAL TRIAL: NCT02734108
Title: Measuring the Effect of a Program of 20 Sessions of Transcranial Direct Current Stimulation With 2 Milli-ampere Targeting the Dorsolateral Prefrontal Cortex on the Symptoms of Anorexia Nervosa: An Open Label Uncontrolled Pilots Study
Brief Title: Transcranial Direct Current Stimulation (tDCS) and Anorexia Nervosa
Acronym: STAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UF 9587; 2015-A00872-47 (Other: ANSM)
Record Dates: First submitted 2016-03-08; First posted 2016-04-12 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Anorexia Nervosa
Keywords: Sever anorexia nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transcranial direct current stimulation (Experimental): 10 patients will be stimulated twice a day for two weeks or 20 sessions. 2 milli ampere stimulation will be applied for 25 min respecting a period of four hours between sessions.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — Anodal transcranial direct current stimulation over the dorsolateral prefrontal cortex

SUMMARY:
Anorexia nervosa is an eating disorder characterized by intense fear of becoming fat despite the obvious thinness and extreme behaviors for weight loss. The result is a massive weight loss and / or pathological thinness. The care of anorexia is difficult and few treatments have proved to be effective in adults.

Transcranial direct current stimulation (tDCS) is a neuromodulation technique that uses an electrical current of low intensity. It allows to modulate the corticospinal excitability: two electrodes, an anode (excitatory) and a cathode (inhibitory), are positioned on the skull according to the region which is desired to influence the operation.

Although tDCS was shown to no noticeable side effects, it is first necessary to assess the feasibility and safety of this technique in these physically frail patients. A recent pilot study suggests the acceptability, safety and efficacy of tDCS program in patients with anorexia nervosa.

Given these preliminary data and the extreme seriousness and vulnerability of patients with resistant anorexia, the investigators want to assess the risk / benefit ratio for the use of this technique in patients suffering from resistant anorexia nervosa. The current data are too preliminary to consider a randomized controlled trial, the investigators hope, initially, replicate the data from this pilot study in a second sample with a more rigorous and comprehensive assessment methodology .

DETAILED DESCRIPTION:
During stimulation, the anode will be placed over the left dorsolateral prefrontal cortex and the cathode on the right dorsolateral prefrontal cortex. Stimulation of 2 milli-Ampere is applied for 25 minutes each session.

20 sessions will be conducted twice a day respecting a period of four hours between sessions.

The tDCS sessions will start maximum 15 days after the inclusion visit.

Two intermediate control visits will be conducted. One after the first week of tDCS, the other immediately after the last session of tDCS.

The main assessment visit will be carried out one month (+/- 5 days) after the last session of tDCS. Finally a reminder visit will be performed 6 months (+/- 3 weeks) after the last session of tDCS to assess the stability over time of the potential effects observed.

ELIGIBILITY:
Inclusion Criteria:

* Present a current anorexia nervosa (according to Diagnostic and Statistical Manual of Mental Disorders (DSM V)) ,severe, for at least 3 years
* Attest to the failure of at least one outpatient treatment conducted by a specialized team (Level 2/3) for the management of patients with eating disorders according to the criteria of French Association for the Development of Specialized Approaches of eating disorders and General Direction of the care
* Have an effective mean of contraception throughout the study
* Being able to understand the nature, purpose and methodology of the study
* Being affiliated to a social security scheme or being the beneficiary of such a scheme.
* Having signed the informed consent

Exclusion Criteria:

* Refusal to participate
* Present a body mass index lower than 13.5
* Present a history of seizures or epilepsy
* Presenting a head injury and / or brain pathology
* Presenting an unstabilized serious physical illness
* Present pregnancy (attested by a blood test Beta-HCG) or breastfeeding
* Present physical disease that may affect cognitive abilities and brain structures (eg HIV infection, multiple sclerosis, lupus, Parkinson's disease, epilepsy, dementia ...)
* Deprived of liberty subject (judicial or administrative decision)
* People protected by law

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-06 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Evolution of the Eating Disorders Examination Questionnaire (EDEq) score | At the baseline and 1 month after the last session of tDCS
  Comparison between the total score of the Eating Disorders Examination Questionnaire (EDEq) 28 days before tDCS program and 28 days after the end of a program of 20 sessions of tDCS with 2 milliampere targeting dorsolateral prefrontal cortex

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by tDCS adverse effect questionnaire | At the end of the first and second week of stimulation
  Evaluate the safety of this program: side effects, early termination of the patient, acceptability
Evolution of depressive symptoms assessed by patients with Beck Depression Inventory (BDI) questionnaire | At the baseline, the end of the first and second week of stimulation, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of mood as an associated symptoms of anorexia nervosa
Evolution of depressive symptoms assessed by the psychiatrist by Montgomery Asberg Depression Rating Scale (MADRS) | At the baseline, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of mood as an associated symptoms of anorexia nervosa
Evolution of mania symptoms assessed by the physician with Young Mania Rating Scale (YMRS) | At the baseline, the end of the first and second week of stimulation, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of mood as an associated symptoms of anorexia nervosa
Evolution of the Exercise Dependence Scale (EDS-R) score | At the baseline, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of physical activity as an associated symptoms of anorexia nervosa
Evolution of the Global Physical Activity Questionnaire (GPAQ) score | At the baseline, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of physical activity as an associated symptoms of anorexia nervosa
Evolution of the Maudsley Obsessive Compulsive Inventory (MOCI) score | At the baseline, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of obsessiveness as an associated symptoms of anorexia nervosa sensitivity
Evolution of the sensitivity to punishment and sensitivity reward questionnaire | At the baseline, 1 month and 6 months after the last session of tDCS
  Evaluate the evolution of reward sensitivity as an associated symptoms of anorexia nervosa sensitivity
Evolution of the neuropsychological performance measured with the National Adult Reading Test (NART) | At the baseline and 1 month after the last session of tDCS
  Evaluate the evolution of neuropsychological performance as an associated symptoms of anorexia nervosa sensitivity
Evolution of the neuropsychological performance measured with the Iowa Gambling Task (IGT) | At the baseline and 1 month after the last session of tDCS
  Evaluate the evolution of neuropsychological performance as an associated symptoms of anorexia nervosa sensitivity
Evolution of the neuropsychological performance measured with the Brixton test | At the baseline and 1 month after the last session of tDCS
  Evaluate the evolution of neuropsychological performance as an associated symptoms of anorexia nervosa sensitivity
Evolution of the neuropsychological performance measured with the Rey-Osterrieth Complex Figure | At the baseline and 1 month after the last session of tDCS
  Evaluate the evolution of neuropsychological performance as an associated symptoms of anorexia nervosa sensitivity
Evolution of the neuropsychological performance measured with the D2 test | At the baseline and 1 month after the last session of tDCS
  Evaluate the evolution of neuropsychological performance as an associated symptoms of anorexia nervosa sensitivity
Evolution of the patient's level of function measured with the Work and Social Adjustment Scale (WSAS) | 6 months
  Evaluate the evolution of the patient's level of function as an associated symptoms of anorexia nervosa sensitivity
Evolution of the patient's level of function measured with the Global Assessment of Functioning (GAF) | 6 months
  Evaluate the evolution of the patient's level of function as an associated symptoms of anorexia nervosa sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien GUILLAUME, MD PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Hopital Lapeyronie, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Strumila R, Thiebaut S, Jaussent I, Seneque M, Attal J, Courtet P, Guillaume S. Safety and efficacy of transcranial direct current stimulation (tDCS) in the treatment of Anorexia Nervosa. The open-label STAR study. Brain Stimul. 2019 Sep-Oct;12(5):1325-1327. doi: 10.1016/j.brs.2019.06.017. Epub 2019 Jun 19. No abstract available. PMID 31239105